CLINICAL TRIAL: NCT02153957
Title: A Randomized Controlled Trial Evaluating an Enhanced Physical Activity Intervention to Improve Cognitive Late Effects in Children Treated With Cranial Radiation for Brain Tumors
Brief Title: Trial Evaluating an Enhanced Physical Activity Intervention to Improve Cognitive Late Effects in Children Treated With Cranial Radiation for Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 140116; 14-C-0116
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-08-20

CONDITIONS: Brain Tumor
Keywords: Exercise; Memory; BDNF; Zamzee; QOL
MeSH Terms: conditions — Brain Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): enhanced PA home intervention group for the first 12 weeks; followed by 12 weeks of PA maintenance on their own.
  Interventions: Behavioral: Physical Activity
- 2 (Active Comparator): usual physical activity (no intervention) for 12 weeks; followed by the enhanced PA home intervention for 12 weeks.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 12 weeks of enhanced physical activity with Zamzee monitor.

SUMMARY:
Background:

- More children with cancer are surviving into adulthood. Some side effects from treatment go away quickly. But some problems may not go away or may only show up months or years later. These problems are called late effects. Late effects can cause difficulties in cognitive functions, such as attention and memory. Physical activity has been found to improve the attention and memory skills of children with Attention Deficit Hyperactivity Disorder (ADHD). Researchers want to see if physical activity can help with these cognitive problems in children with brain tumors.

Objectives:

- To see if physical activity can improve cognitive functions in children who had radiation therapy for a brain tumor.

Eligibility:

- Children ages 8 17 who had radiation for a brain tumor at least 2 years ago. They must have access to a computer.

Design:

* Participants will be screened with height, weight, and medical history. They will answer questions about daily physical activities. Their heart will be checked.
* Participants will go to the clinic for 2 days. They will have a fitness exam and tests about attention, memory, and concentration. They will have blood taken and answer questions. Parents will also answer questions.
* Participants will be put into 2 groups. For the first 12 weeks, the intervention group will follow a physical activity program. The control group will do their usual physical activities.
* For the second 12 weeks, the control group will follow the physical activity program. The intervention group will continue the activities on their own. All groups will track their physical activity with an activity monitor and computer.
* Participants will have a follow-up visit at the clinic after each session. They will repeat some of the tests listed above.
* The study lasts 24 weeks plus the two follow-up visits. Participants can keep their activity monitor.

DETAILED DESCRIPTION:
BACKGROUND:

* Children treated with cranial radiation therapy (CRT) for brain tumors are at high risk for developing neurocognitive late effects consisting of significant declines in overall IQ and specific cognitive impairments, particularly in attention, memory, and processing speed. Academic functioning, daily activities, and quality of life (QOL) also are impacted, and children often require special educational services.
* Despite adaptations in radiation therapy (delay of radiation, reduced dose, specialized techniques), cognitive deficits still develop. Interventions targeting cognitive rehabilitation are limited yet sorely needed.
* A potential and novel intervention for cognitive rehabilitation that has not been explored in children with cancer involves physical activity (PA). Compelling evidence from both human and animal studies indicates that PA affects the same brain mechanisms and cognitive functions damaged by CRT and chemotherapy.
* Previous PA intervention studies in children with cancer have been found to be feasible, safe, and beneficial to health but have not examined cognition outcomes. Therefore, we will conduct a randomized controlled trial to evaluate the effects of PA on the cognitive functioning of children treated with CRT for brain tumors. In addition, we will enhance the intervention by combining it with Acceptance and Commitment Therapy (ACT) techniques to maximize participants' motivation to engage in PA.
* The immediate intervention group (the intervention group ) will engage in the enhanced PA intervention program for the first 12 weeks followed by 12 weeks of PA maintenance on their own, while the delayed intervention control group (the control group ) will engage in their usual physical activity for the first 12 weeks followed by the enhanced PA intervention program for the second 12 weeks.

OBJECTIVES:

-To assess the effects of a 12-week enhanced physical activity (PA) home intervention on visual memory (CogState One Card Learning Accuracy score) in children treated with CRT for brain tumors compared to a control group engaged in usual physical activity during the first 12 weeks.

ELIGIBILITY:

* Children ages 8 - 18 years previously diagnosed with a brain tumor in childhood who are at least 1 year post-completion of CRT and who are not on an active anti-tumor treatment will be eligible.
* Children should have reported or documented cognitive difficulties in attention, learning and memory, or processing speed per the child s parent or legal guardian.

DESIGN:

-In this prospective randomized controlled trial. Children will be randomized to one of two groups: Group 1 (n=30): The immediate intervention group (the intervention group ) will participate in the enhanced PA home intervention group for the first 12 weeks; followed by 12 weeks of PA maintenance on their own.

Group 2 (n=30): The delayed intervention control group (the control group ) will engage in their usual physical activity (no intervention) for 12 weeks; followed by the enhanced PA home intervention for 12 weeks.

* Neurobehavioral, circulating growth factors, and cardiorespiratory evaluations will be conducted at baseline (T0) and after the first 12 weeks at home (T2) in both the intervention and control groups. The acute effects of the in-lab PA will be assessed immediately following the baseline treadmill fitness test (T1) using selected cognitive measures in both groups. PA for both groups will be measured throughout the period at home via activity monitors.
* After the completion of the first 12 week period at home and the follow-up evaluations (T2), the intervention group will be asked to maintain their PA levels on their own for the next 12 weeks while the control group will participate in the enhanced PA intervention at home for 12 weeks. A final cognitive evaluation will be conducted in both groups after the completion of the second 12- week period (T3). The primary outcome measure is the Cogstate One Card Learning Accuracy Score. The effects of PA on other neurobehavioral outcomes and circulating growth factors also will be examined.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Children ages 8 - 18 years of age, diagnosed with brain tumor in childhood.
  2. Must be at least 1 year post completion of radiation therapy to the brain or brain and spine.
  3. Must be off anti-neoplastic therapy for at least 2 weeks and all therapy-related toxicities should return to baseline or less than or equal to Grade 1 if previously nonexistent.
  4. Have parent-reported or documented difficulties in attention, processing speed, memory, or learning as assessed by the screening questions (a score of at least 3 on any one of the 4 questions or the participant having greater than or equal to 1/2 SD decline in test scores, scores < 85, or special education services or accommodations).
  5. Must have a parent or legal guardian willing to complete the parent proxy behavioral questionnaires and help their child participate in the study procedures at home.
  6. Ability to read and understand the English language.
  7. Have regular access to a computer a tablet, or a smartphone (the device must have either a USB port or Bluetooth with internet capability).
  8. Must be willing to register online and install the software to use an age-appropriate activity monitor and website/app which will include sharing some personal identifiable information, to allow the participant to track their physical activity.
  9. Ability of subject or parent/guardian to understand and willingness to sign a written informed consent document.

PARENT OR GURADIAN OF PARTICIPATING SUBJECT:

1. Parent or Guardian of participating subject
2. Ability to understand and willingness to sign a written informed consent document
3. Ability to read and understand the English language.

EXCLUSION CRITERIA

1. A child with diffuse intrinsic pontine glioma (DIPG) or recurrent high grade brain tumors will be excluded due to the poor prognosis, making participation for the length of this study difficult.
2. Significant medical problems, such as severe uncontrolled illnesses, or physical impairments that prohibit the child from exercising at moderate to vigorous levels based on the clinical judgment of the examining physician or nurse practitioner.
3. Currently engaging in > 3 hours of moderate to vigorous physical activity per week, as reported in the exercise screening questions completed at the pre-study screening evaluation.
4. Significant cognitive, behavioral, or emotional impairments as judged by an investigator that would prevent the child from understanding or completing the intervention or assessment measures.
5. A child has plans to start a new treatment for attention/memory problems in the next 3 months.
6. Currently on or planning to begin active neoplastic therapy, as the side effects may significantly impair ability to participate in physical activity.
7. Unable or unwilling to travel to NIH or DFCI/BCH for the evaluations.
8. History of medical non-compliance or difficulty completing previous required study tasks or visits that suggest the participant would not follow through with the home study procedures.

PARENT OR GUARDIAN EXCLUSION CRITERIA:

1. Parent or guardian of an ineligible subject

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 weeks
  Efficacy of 12-weeks PA on visual memory

SECONDARY OUTCOMES:
feasibility | 4 years
  To assess the feasibility of various components of the intervention (e.g., ACT sessions, PA monitors) based on the post-study questionnaire/interview and explore relationships between the use of these components and physical activity outcomes
examine test scores pre- to post-intervention | 24 weeks
  examine test scores pre- to post-intervention
effects of lab treadmill on neurobehavioral functioning | 2 days
  effects of lab treadmill on neurobehavorial functioning
effects of 12wk PA on fatigue, sleep and QOL | 24 weeks
  effects of 12wk PA on fatigue, sleep, and QOL
effects of 12wk PA on cognitive functions | 24 weeks
  effects of 12wk PA on cognitive functions
compare cognitive test scores between groups | 12 weeks
  compare cognitive test scores between groups

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Wolters, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Naylor AS, Bull C, Nilsson MK, Zhu C, Bjork-Eriksson T, Eriksson PS, Blomgren K, Kuhn HG. Voluntary running rescues adult hippocampal neurogenesis after irradiation of the young mouse brain. Proc Natl Acad Sci U S A. 2008 Sep 23;105(38):14632-7. doi: 10.1073/pnas.0711128105. Epub 2008 Sep 2. PMID 18765809
- [Background] Gapin JI, Labban JD, Etnier JL. The effects of physical activity on attention deficit hyperactivity disorder symptoms: the evidence. Prev Med. 2011 Jun;52 Suppl 1:S70-4. doi: 10.1016/j.ypmed.2011.01.022. Epub 2011 Jan 31. PMID 21281664
- [Background] Butryn ML, Forman E, Hoffman K, Shaw J, Juarascio A. A pilot study of acceptance and commitment therapy for promotion of physical activity. J Phys Act Health. 2011 May;8(4):516-22. doi: 10.1123/jpah.8.4.516. PMID 21597124
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0116.html